CLINICAL TRIAL: NCT02610530
Title: Efficacy of Surgical Intervention for the Treatment of Diabetes Mellitus Type 2 in Overweight Non-responders in Comparison With Conventional Nonsurgical Medical Treatment
Brief Title: Surgical Intervention for the Treatment of Diabetes in Overweight Non-responders-1
Acronym: SIT-DOWN-1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Turkish Metabolic Surgery Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/S01
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Overweight; Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; metabolic surgery; medical treatment
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2 | interventions — Hypoglycemic Agents; Insulin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-Surgery: Overweight diabetic, type 2 diabetes diagnosis longer than 3 years; BMI:25-29.9 kg/m2 who have been on medical treatment for glycemic control.
  Interventions: Other: Medical Treatment
- Surgery-A: Overweight diabetic, type 2 diabetes diagnosis longer than 3 years; BMI:25-29.9 kg/m2. who underwent sleeve gastrectomy with ileal transposition
  Interventions: Procedure: Sleeve Gastrectomy with Ileal Transposition
- Surgery-B: Overweight diabetic, type 2 diabetes diagnosis longer than 3 years; BMI:25-29.9 kg/m2. who underwent sleeve gastrectomy with transit bipartition
  Interventions: Procedure: Sleeve Gastrectomy with Transit Bipartition

INTERVENTIONS:
Procedure: Sleeve Gastrectomy with Ileal Transposition — Type 2 diabetic patients who underwent ileal transposition surgery within the last 2 years.
  Groups: Surgery-A
Procedure: Sleeve Gastrectomy with Transit Bipartition — Type 2 diabetic patients who underwent transit bipartition surgery within the last 2 years.
  Groups: Surgery-B
Other: Medical Treatment — Conventional Non-Surgical Treatment for Glycemic Control group consisted of patients who did not undergo any kind of surgery, and are on medical treatment for type 2 diabetes.
  Other Names: Oral antidiabetics and / or insulin
  Groups: Non-Surgery

SUMMARY:
The SIT-DOWN study is a single centered retrospective study in which a total of 90 (ninety) participants who are overweight (BMI: 25-29.9 kg/m2) and have type 2 diabetes mellitus (T2DM) will be evaluated for the efficacy of surgical intervention in comparison with medical treatment. Primary endpoint of the study will be the change in glycemic regulation by the end of 12 months.

DETAILED DESCRIPTION:
Use of bariatric/metabolic surgery has conventionally been reserved for those whose body-mass index (BMI) is 35 kg/m2 or greater. Trials in these morbidly obese patients confirmed the benefits in terms of weight loss and provide evidence that surgery can result in remission of diabetes, and as a result lead to improvement in cardiovascular risk factors. Within the light of these data, there appear to be a shift towards lower BMI, with many advocating it as a reasonable option for diabetics with a lower BMI (<30) who have failed other attempts of medical treatment. But this approach is limited because of lack of data on the effects of surgical outcomes in this group of patients which is the main rationale for this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Overweight, type 2 diabetic: Type 2 diabetes diagnosis longer than 3 years; BMI= 25-29.9 kg/m2
* Participants with baseline HbA1c ≥ % 7.5, not achieved HbA1c < % 7.3 at 3 months on therapy
* Absence of co-morbidities (neuropathy, retinopathy, cardiovascular disease, stroke events or lower extremity amputation).

Exclusion Criteria:

* Liver cirrhosis, severe renal failure, collagen diseases, severe endocrinopathies, blindness.
* Heart failure, acute myocardial infarction, stroke or transient ischemic attack, unstable angina pectoris.
* History of malignancy or malignant neoplasm in place, severe inflammatory complications, neurological or cardiovascular in act.
* Pregnancy
* Any conditions that at the discretion of the head of the study can represent risk to the participant or could affect the protocol results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight, type 2 diabetic: Type 2 diabetes diagnosis longer than 3 years; BMI= 25-29.9 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in glycated hemoglobin (HbA1c) | 1 year
  Complete diabetic remission (HbA1c < 6%) and partial diabetic remission (HbA1c= 6-6.5%) without medication.

SECONDARY OUTCOMES:
Hypertension Control | 1 year
  Systolic blood pressure (BP) <130 mm Hg and diastolic BP <80 mm Hg, without medication.
Change in LDL (low-density lipoprotein) Cholesterol | 1 year
  <100 mg/dL, without medication.
Change in HDL (high-density lipoprotein) Cholesterol | 1 year
  >40 mg/dL, without medication.
Change in Triglycerides | 1 year
  <150 mg/dL, without medication.
Weight Control | 1 year
  Amount of weight loss in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Celik, MD, Principal Investigator — Turkish Metabolic Surgery Foundation

REFERENCES:
- [Background] DePaula AL, Macedo AL, Schraibman V, Mota BR, Vencio S. Hormonal evaluation following laparoscopic treatment of type 2 diabetes mellitus patients with BMI 20-34. Surg Endosc. 2009 Aug;23(8):1724-32. doi: 10.1007/s00464-008-0168-6. Epub 2008 Oct 2. PMID 18830747
- [Background] Kashyap SR, Daud S, Kelly KR, Gastaldelli A, Win H, Brethauer S, Kirwan JP, Schauer PR. Acute effects of gastric bypass versus gastric restrictive surgery on beta-cell function and insulinotropic hormones in severely obese patients with type 2 diabetes. Int J Obes (Lond). 2010 Mar;34(3):462-71. doi: 10.1038/ijo.2009.254. Epub 2009 Dec 22. PMID 20029383
- [Background] Finelli C, Padula MC, Martelli G, Tarantino G. Could the improvement of obesity-related co-morbidities depend on modified gut hormones secretion? World J Gastroenterol. 2014 Nov 28;20(44):16649-64. doi: 10.3748/wjg.v20.i44.16649. PMID 25469034
- [Background] Kashyap SR, Bhatt DL, Wolski K, Watanabe RM, Abdul-Ghani M, Abood B, Pothier CE, Brethauer S, Nissen S, Gupta M, Kirwan JP, Schauer PR. Metabolic effects of bariatric surgery in patients with moderate obesity and type 2 diabetes: analysis of a randomized control trial comparing surgery with intensive medical treatment. Diabetes Care. 2013 Aug;36(8):2175-82. doi: 10.2337/dc12-1596. Epub 2013 Feb 25. PMID 23439632
- [Background] Santoro S. From Bariatric to Pure Metabolic Surgery: New Concepts on the Rise. Ann Surg. 2015 Aug;262(2):e79-80. doi: 10.1097/SLA.0000000000000590. No abstract available. PMID 24646534
- [Background] Celik A, Ugale S. Functional restriction and a new balance between proximal and distal gut: the tools of the real metabolic surgery. Obes Surg. 2014 Oct;24(10):1742-3. doi: 10.1007/s11695-014-1368-x. No abstract available. PMID 25027983
- [Background] Santoro S, Castro LC, Velhote MC, Malzoni CE, Klajner S, Castro LP, Lacombe A, Santo MA. Sleeve gastrectomy with transit bipartition: a potent intervention for metabolic syndrome and obesity. Ann Surg. 2012 Jul;256(1):104-10. doi: 10.1097/SLA.0b013e31825370c0. PMID 22609843
- [Background] De Paula AL, Stival AR, Halpern A, DePaula CC, Mari A, Muscelli E, Vencio S, Ferrannini E. Improvement in insulin sensitivity and beta-cell function following ileal interposition with sleeve gastrectomy in type 2 diabetic patients: potential mechanisms. J Gastrointest Surg. 2011 Aug;15(8):1344-53. doi: 10.1007/s11605-011-1550-6. Epub 2011 May 10. PMID 21557013
- [Background] De Paula AL, Stival AR, Macedo A, Ribamar J, Mancini M, Halpern A, Vencio S. Prospective randomized controlled trial comparing 2 versions of laparoscopic ileal interposition associated with sleeve gastrectomy for patients with type 2 diabetes with BMI 21-34 kg/m(2). Surg Obes Relat Dis. 2010 May-Jun;6(3):296-304. doi: 10.1016/j.soard.2009.10.005. Epub 2009 Nov 10. PMID 20096647